CLINICAL TRIAL: NCT06244810
Title: Comparison of Two Types of Lingual Fixed Retainer (Metal and Fiber)Fabricated by Using (CAD\CAM)Technique
Brief Title: Comparison of Two Types of Lingual Fixed Retainer Fabricated
Acronym: malocclusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hama University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hama University -Dentistry
Record Dates: First submitted 2024-01-22; First posted 2024-02-06 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Malocclusion, Angle's Class
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lingual retainer made of fiber made using cad cam Technique (Experimental): lingual retainer made of fiber manufactured using CAD-CAM technique applied to the lingual surfaces of the mandibular incisors and evaluated every month over a period of 6 months.
  Interventions: Device: Lingual retainer from Fiber
- lingual retainer made of metal made using cad cam Technique (Experimental): lingual retainer made of metal manufactured using CAD-CAM technique applied to the lingual surfaces of the mandibular incisors and evaluated every month over a period of 6 months
  Interventions: Device: Lingual retainer from metal
- Traditional lingual retainer made of braided stainless steel wire (Experimental): lingual retainer made of braided stainless steel wire applied to the lingual surfaces of the mandibular incisors and evaluated every month over a period of 6 months.
  Interventions: Device: Traditional retianer from braided

INTERVENTIONS:
Device: Lingual retainer from Fiber — lingual retainer manufactured from fiber using CAD-CAM technique applied to the lingual surfaces of the mandibular incisors and evaluated every month over a period of 6 months.
  Arms: lingual retainer made of fiber made using cad cam Technique
Device: Lingual retainer from metal — lingual retainer manufactured from metal using CAD-CAM technique applied to the lingual surfaces of the mandibular incisors and evaluated every month over a period of 6 months.
  Arms: lingual retainer made of metal made using cad cam Technique
Device: Traditional retianer from braided — lingual retainer manufactured using traditional technique from stainless steel applied to the lingual surfaces of the mandibular incisors and evaluated every month over a period of 6 months.
  Arms: Traditional lingual retainer made of braided stainless steel wire

SUMMARY:
This study includes patients who have had previous orthodontic treatments (without tooth extraction) and who have good alignment of their lower incisors. Investigators will compare two types of lingual retainers made with CAD-CAM

DETAILED DESCRIPTION:
This study includes patients who have had previous orthodontic treatments (without tooth extraction) and who have good alignment of their lower incisors. Investigator will compare two types of lingual retainers made with CAD-CAM by comparing them with the traditional lingual retainers according to the following groups:

1. Patients will be apply to them a lingual retainer made of fibers manufactured using CAD-CAM technology
2. Patients will be apply to them a lingual retainer made of metal made using CAD-CAM technology
3. Patients will be apply to them a conventional lingual retainer made of braided stainless steel wire (control group)

ELIGIBILITY:
Inclusion Criteria:

* Patients with mixed dentition at age 14-24 years. They have a good alignment of the lower incisors.- Have good oral and periodontal health.-

Exclusion Criteria:

Patients who have a deep bite Patients who have previously used retainer Patients with poor oral care

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-03-09 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Bacterial plaque indicator | 6 months
  the amount of plaque on the gingival edge on the tooth surface is determined by using a probe. This indicator does not need to color the plaque. This indicator is taken for all teeth monthly over a period of 6 months
Patient Acceptance Assessment: | 6 months
  Patient acceptance will be evaluated according to a set of questions presented in a questionnaire sheet for each patient in the hospital
  Each period of the review where patient acceptance was recorded in three aspects:
  1. Speech: The extent of the effect of the affixed fixative on the patient's comfort with speech will be recorded in each follow-up period in the event that there is no difficulty in speaking or there is difficulty in speaking.
     Is there a proven effect on speech? )Yes No(
  2. Oral Care Procedures: The patient's ability to perform oral care procedures will be recorded In my case, the ease and difficulty of doing oral care procedures. How easy is it for you to perform oral care procedures? (easy / hard)

CONTACTS AND LOCATIONS:
Overall Officials: Manar A Warrar, MSc, Principal Investigator — Hama University-Syrian Arab Republic; Rabab Alsabbagh, Professor, Study Chair — Professor of Orthodontics, University of Hama Dental School, Hama, Syria.
Locations (1):
- FADI Alhaji JNAID, Damascus, None Selected, Syria

IPD SHARING:
Plan to Share IPD: No